CLINICAL TRIAL: NCT04197674
Title: China Q Cohort Study: an Extended Follow-up Study of PD vs. HD Randomized Trial
Brief Title: China Q Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xue Qing Yu, Professor, Sun Yat-sen University
Other Study IDs: China Q Cohort
Record Dates: First submitted 2019-11-29; First posted 2019-12-13 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: End Stage Renal Disease on Dialysis; Peritoneal Dialysis; Hemodialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Peritoneal dialysis group: Patients who randomized to peritoneal dialysis
  Interventions: Other: Dialysis modality
- Hemodialysis group: Patients who randomized to conventional in-center hemodialysis
  Interventions: Other: Dialysis modality

INTERVENTIONS:
Other: Dialysis modality — This is a observational cohort study, and there is no intervention for all participants. Our aim is to evaluate dialysis modality (PD and HD) on patient survival

SUMMARY:
The burden of end-stage kidney disease (ESKD) is increasing worldwide. Although kidney transplantation is the most cost-effective renal replacement therapy, dialysis is still the main way to treat ESRD patients due to the limited kidney donor, with approximately 89% of such dialysis patients receive hemodialysis (HD) and the remainder receive peritoneal dialysis (PD). This distribution of dialysis modality, however, varies widely by health jurisdiction. For instance, more than 97% of dialysis patients are treated with HD in Japan, but more than 50% treated with PD in Mexico. Evidence comparing the two modalities suggests that mortality risks may be comparable, but all evidence come from observational study and there is no randomized controlled trial to compare patient survival between PD and HD due to patients enrollment issue.More importantly, for most health care systems, such as United States, United Kingdom, Australia, Indonesia and China, PD is less expensive than HD. It is possible, then, that a greater global utilization of PD might improve access to renal replacement therapy in less advanced economies.

The investigators have conducted a prospective, randomized, parallel, open-label, multi-center, non-inferiority trial to evaluate health-related quality of life (HRQoL) with PD versus conventional in-center HD in incident ESKD patients. A total of 1082 ESKD patients were randomly assigned to PD or conventional in-center HD, and 235 patients enrolled in stage 1 with complete measures of the "Burden of Kidney Disease" at both baseline and 48 weeks and 668 patients enrolled in stage 2 were included in analysis. However, this trial was designed to evaluate quality of life between PD and HD and all patients were follow-up 48 weeks. Therefore, in this observational cohort study, the investigators will perform extended follow-up for participants including in analysis . Our primary objective is to evaluate the association of dialysis modality (PD and HD) with all-cause mortality in ESKD patients. The investigators also explore the impact of PD and HD on major cardiovascular event composite (MACE), a composite outcome of MACE and all-cause death, hospitalized myocardial infarction, hospitalized stroke and hospitalized heart failure, healthy utility, dialysis cost, activity of daily living, and changes of RRF, hemoglobin, and other biochemical parameters.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥ 18 years old) peritoneal dialysis or in-center hemodialysis patient who have been recruited in previous China Q study and who enrolled in SURinD study with complete measures of the "Burden of Kidney Disease" at both baseline and 48 weeks.
* Will and able to provide the informed consent form (ICF).

Exclusion Criteria:

* Patients have stopped dialysis due to kidney function recovery or kidney transplantation.
* Patients refuse to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: End stage kidney disease patients who randomly assigned to receive peritoneal dialysis and conventional in-center hemodialysis
Sampling Method: Probability Sample
Enrollment: 903 (Estimated)
Dates: Start 2020-01-21 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants died due to any cause | From the first day receiving assigned treatment to the end of 3rd year follow-up
  Patients died due to any cause

SECONDARY OUTCOMES:
Number of Participants with major cardiovascular event composite (MACE) | From the first day receiving assigned treatment to the end of 3rd year follow-up
  MACE defined as defined as the first occurrence of myocardial infarction, ischemic stroke or death from cardiovascular causes
Number of Participants with composite outcome of MACE and all-cause death | From the first day receiving assigned treatment to the end of 3rd year follow-up
  Patients experience cardiovascular events and death.
Number of Participants with hospitalized myocardial infarction, stroke and heart failure | From the first day receiving assigned treatment to the end of 3rd year follow-up
  Patients were hospitalized due to myocardial infarction, stroke and heart failure.
Healthy utility | From the first day receiving assigned treatment to the end of 3rd year follow-up
  Healthy utility was assessed by Kidney Disease Quality of Life-Short Form (KDQoL-SF™, version 1.3) questionnaire domain of General health, with a range of 1 to 100 and higher value indicates better healthy utility
Rate of difference in dialysis cost between PD and HD | From the first day receiving assigned treatment to the end of 3rd year follow-up
  Dialysis cost is evaluated by budget impact model which is developed by Baxter Healthcare Corporation and is a excel based calculator with higher value indicates higher cost
Changes of activity of daily living | From the first day receiving assigned treatment to the end of 3rd year follow-up
  Activity of daily living assessed using Activrty Daily Living (ADL) scale, with a range of 14 to 56 and a score < 14 indicates independent daily living and a higher score indicates serious dependent daily living.
Changes of residual renal function | From the first day receiving assigned treatment to the end of 3rd year follow-up
  Residual renal function was evaluated using 24h urine volume and the unit is ml.
Changes of hemoglobin | From the first day receiving assigned treatment to the end of 3rd year follow-up
  The unit of hemoglobin is g/L.
Changes of serum phosphors | From the first day receiving assigned treatment to the end of 3rd year follow-up
  The unit of serum phosphors is mmol/L.
Changes of serum albumin | From the first day receiving assigned treatment to the end of 3rd year follow-up
  The unit of serum albumin is g/L.

CONTACTS AND LOCATIONS:
Overall Officials: Xueqing Yu, Principal Investigator — yuxq@mail.sysu.edu.cn
Locations (1):
- The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
Data share plan will decided before submit manuscript to journal.

REFERENCES:
- [Derived] Ethier I, Hayat A, Pei J, Hawley CM, Johnson DW, Francis RS, Wong G, Craig JC, Viecelli AK, Htay H, Ng S, Leibowitz S, Cho Y. Peritoneal dialysis versus haemodialysis for people commencing dialysis. Cochrane Database Syst Rev. 2024 Jun 20;6(6):CD013800. doi: 10.1002/14651858.CD013800.pub2. PMID 38899545